CLINICAL TRIAL: NCT02310815
Title: ReSure Sealant Post-Approval Study: A Registry Evaluation of ReSure Sealant for Specified Adverse Ocular Events After Sealing Corneal Incisions in Patients Undergoing Clear Corneal Cataract Surgery
Brief Title: ReSure Sealant Post Approval Study
Acronym: Clinical PAS
Status: Completed | Type: Observational
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OTX-13-003
Record Dates: First submitted 2014-12-03; First posted 2014-12-08 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Adverse Events

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ReSure Sealant

SUMMARY:
This is a prospective multicenter observational post-approval registry study that will collect post-approval data relative to the incidence of pre-specified Adverse Ocular Events for cataract surgery patients treated with the FDA-approved ReSure Sealant when used by a broad group of physicians under commercial use conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a cataract and is expected to undergo clear corneal cataract surgery with intraocular lens placement

Exclusion Criteria:

* ReSure Sealant is not applied to the operative eye

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with ReSure Sealant following cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 626 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Anterior chamber cells greater than level 1+ persisting at Visit 2 (≥ Day 20) | Post operative days 20 to 40
Hypotony (≤ 5 mmHg) | Post operative days 20 to 40
Ocular discomfort | Post operative days 20 to 40
  Ocular Comfort Index score greater than 51.7 or a within-person increase from baseline of greater than 37.8
Surgical reintervention | Post operative days 20 to 40
  Surgical reintervention for management of a wound leak - Yes or No